CLINICAL TRIAL: NCT00731380
Title: Phase I Trial of ABI-007 (Abraxane) Plus Cisplatin Plus 5-Fluorouracil (APF) as Induction Chemotherapy Followed by Concurrent Chemoradiotherapy in Patients With Locally Advanced Squamous Cell Cancers of the Head and Neck (HNSCC)
Brief Title: A Phase I Trial of Abraxane, Cisplatin and 5-Fluorouracil Along With Chemoradiotherapy in Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APF-001
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Cancer
Keywords: Abraxane; Head and Neck Cancer; Determine; Maximum; Tolerated dose; ABI-007; Combination; Cisplatin; 5-Fluorouracil; Patients
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-007 escalation; then radiation + AUC (Experimental): Dose escalation beginning with ABI-007 75 mg/m2 day 1 + day 8, Cisplatin 100 mg/m2 day 1, 5-FU 1000 mg/m2/d continuous infusion x 96 hours on day 1-4, for 3 weeks x 3 cycles. Followed by Concurrent weekly Carboplatin (AUC 1.5) with radiotherapy for 7 weeks. Carboplatin should be given on Monday or Tuesday of each week, if possible.
  Interventions: Drug: ABI-007

INTERVENTIONS:
Drug: ABI-007 — Dose escalation beginning with ABI-007 75 mg/m2 day 1 + day 8, Cisplatin 100 mg/m2 day 1, 5-Fluorouracil (5-FU) 1000 mg/m2/d continuous infusion x 96 hours on day 1-4, for 3 weeks x 3 cycles. Followed by Concurrent weekly Carboplatin (AUC 1.5) with radiotherapy for 7 weeks. Carboplatin should be given on Monday or Tuesday of each week, if possible.
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to determine the highest dose of a ABI-007 that can be given with cisplatin and 5-fluorouracil without causing intolerable side effects in patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck (HNSCC) is the 9th most common malignancy diagnosed in Canadians. In the year 2007, there was an estimated 4,350 new cases diagnosed in Canada, with approximately 1,600 deaths attributable to HNSCC[Canadian Cancer Statistics 2007]. In the United States there is an annual incidence of approximately 40,000 newly diagnosed cases of head and neck cancer [US Cancer Statistics 2006]. Primary treatment for newly diagnosed localized (stage I-II) HNSCC is surgery and/or radiotherapy. The majority of patients (70%) however present with locally advanced HNSCC (Stage III or IV). Treatment of locally advanced HNSCC generally consists of either concurrent chemotherapy and radiation or surgical resection followed by adjuvant radiation or adjuvant concurrent chemotherapy and radiation. Unfortunately despite aggressive treatment with combined modality therapies approximately 40-50% of cases recur, with the majority recurring at the primary site and/or regional nodes. Except for a small minority of patients in whom salvage surgery or radiotherapy can be delivered, the prognosis for the majority of these patients is poor and further treatment is generally considered palliative.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx. Histological or cytological confirmation is required. The disease must be considered to be potentially curable by combined chemoradiation. Patients with nasopharynx, paranasal sinus, skin or unknown primary sites are not eligible.
2. Non-metastatic, stage III or IV disease (UICC/AJCC classification, 6th edition)
3. Age ≥ 18.
4. ECOG performance status of 0 or 1.
5. Patients must have adequate hematological function:

   * absolute granulocyte count > 1.5 x 109/L
   * platelet count >100 x 109/L
   * hemoglobin > 90 g/L
6. Must have adequate renal and hepatic function:

   * serum bilirubin < 1.5x UNL and AST/ALT <2.5x UNL
   * serum creatinine < 1.25 x UNL or a calculated creatinine clearance of > 60 ml/min
7. Signed written consent.
8. Availability for follow-up for up after treatment.
9. The patient is fertile and is aware of the risk of becoming pregnant or fathering children and will use adequate contraception (oral contraception, IUD, diaphragm and spermicide or male condom and spermicide) throughout therapy and for at least 3 months after therapy.
10. Life expectancy greater than 6 months

Exclusion Criteria:

1. Significant inter-current illness that will interfere with the chemotherapy or radiation therapy during the trial such as HIV infection, cardiac insufficiency, pulmonary compromise, active significant alcohol abuse, uncontrolled psychotic disorder, active infection or febrile illness.
2. Any history of myocardial infarction, any history of ventricular arrhythmias, angina or active coronary heart disease within 6 months. Significant cardiac disease resulting in an inability to tolerate the intravenous fluid load as required for administration of cisplatin.
3. Evidence of distant metastases.
4. Symptomatic peripheral neuropathy ≥ grade 1 by CTCAE v.3 criteria.
5. Clinically significant sensorineural hearing impairment which may be exacerbated by cisplatin (audiometric abnormalities without corresponding clinical deafness will not be grounds for exclusion)
6. Weight loss greater than 20% of usual body weight in the 3 months preceding trial entry.
7. High risk for poor compliance with therapy or follow-up as assessed by investigator.
8. Pregnant or lactating women.
9. Prior radiation therapy to greater than 30% of the bone marrow
10. Prior experimental therapy for cancer within 30 days of entering the trial.
11. Prior radiation for head and neck cancer.
12. Prior systemic chemotherapy for cancer.
13. Patients with prior cancers, except: those diagnosed more than five years ago with no evidence of disease recurrence and a clinical expectation of recurrence of less than 5%; or successfully treated non-melanoma skin cancer; or carcinoma in situ of the cervix. However, any patient with previous invasive breast cancer, prostate cancer or melanoma is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of ABI-007 with Cisplatin and 5-Fluorouracil (APF) | two years

SECONDARY OUTCOMES:
safety and tolerability profiles for ABI-007 | two years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Loong HH, Winquist E, Waldron J, Chen EX, Kim J, Palma D, Read N, Razak AR, Diaz-Padilla I, Chan K, Bayley A, Hossain M, Wang L, Chin S, Siu LL, Hope A. Phase 1 study of nab-paclitaxel, cisplatin and 5-fluorouracil as induction chemotherapy followed by concurrent chemoradiotherapy in locoregionally advanced squamous cell carcinoma of the oropharynx. Eur J Cancer. 2014 Sep;50(13):2263-70. doi: 10.1016/j.ejca.2014.05.021. Epub 2014 Jun 19. PMID 24953566